CLINICAL TRIAL: NCT00840658
Title: Epidemiologic Study on Changing HIV Risks Among FSW-IDUs on the Mexico-US Border
Brief Title: Behavioral Intervention to Reduce Sexual and Injection Risks Among Female Sex Workers Who Also Inject Drugs in Mexico
Acronym: FSW-IDU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steffanie Strathdee (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, San Diego (Other); ISSESALUD (Unknown); Universidad Autonoma de Ciudad Juarez (Other); Northeastern University (Other); San Diego State University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Steffanie Strathdee, Principal Investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: DESPR R01DA023877; R01DA023877 (NIH); 5R01DA023877-02 (NIH); NCT01719939 (obsolete NCT alias)
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Results first posted 2012-09-18 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Injection drug users; Female sex workers; STIs; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Drug Interactions; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Placebo Comparator): Didactic safer injection & sexual activity education: In each city, 75 women will participate in a 60 minute lecture-format presentation and printed materials on safer sex and safer injection based on CDC guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). In this component, there will be no theory-driven active skill building elements oriented towards safer sex or safer injection.
  Interventions: Behavioral: Lecture-format presentation
- Group B (Active Comparator): Interactive injection risk intervention and didactic safer sex education: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] counseling session. This one-on-one intervention incorporates elements of motivational interviewing (MI) and principles of Social Cognitive Theory and Theory of Reasoned Action (SCT/TRA) to address the context of unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared. In addition, participants will be provided a lecture-format presentation on safer sex. However, in this component, there will be no theory-driven active skill building elements oriented towards safer sex.
  Interventions: Behavioral: Interactive Injection Risk Intervention
- Group C (Active Comparator): Interactive sexual risk intervention and didactic safer injection education: In each city, 75 women will participate in the 60 minute "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one on one intervention incorporates elements of MI and principles of Social Cognitive Theory and Theory of Reasoned Action (SCT/TRA) to address the context of unsafe sex and condom use with clients. In addition, participants will be provided a lecture format presentation on safer injection sharing. However, in this component, there will be no theory-driven active skill building elements oriented towards safer injection behavior.
  Interventions: Behavioral: Interactive Sexual Risk Intervention
- Group D (Experimental): Interactive injection and sexual risk intervention: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] and "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one-on-one intervention incorporates elements of MI and principles of Social Cognitive Theory and Theory of Reasoned Action (SCT/TRA) to address the context of both, a) unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared; and b) unsafe sex and condom use with clients, and associated risks (e.g., HIV (Human Immuno-deficiency Virus), STIs (Sexually Transmitted Infections), pregnancy).
  Interventions: Behavioral: Interactive injection and sexual risk intervention

INTERVENTIONS:
Behavioral: Interactive injection and sexual risk intervention — This is a one-on-one intervention that incorporates elements of motivational interviewing (MI) and principles of Social Cognitive Theory (SCT) and Theory of Reasoned Action (TRA) to address the context of both, a) unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared; and b) unsafe sex and condom use with clients, and associated risks (e.g., HIV (Human Immuno-deficiency Virus), STIs (Sexually Transmitted Infections), pregnancy).
  Other Names: Motivational Interviewing
  Arms: Group D
Behavioral: Interactive Sexual Risk Intervention — This is a one-on-one intervention that incorporates elements of motivational interviewing (MI) and principles of Social Cognitive Theory (SCT) and Theory of Reasoned Action (TRA) to address the context of unsafe sex and condom use with clients, and associated risks (e.g., HIV (Human Immuno-deficiency Virus), STIs (Sexually Transmitted Infections), pregnancy).
  Other Names: Motivational interviewing
  Arms: Group C
Behavioral: Interactive Injection Risk Intervention — This is a one-on-one intervention that incorporates elements of motivational interviewing (MI) and principles of Social Cognitive Theory (SCT) and Theory of Reasoned Action (TRA) to address the context of unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared.
  Other Names: Motivational interviewing
  Arms: Group B
Behavioral: Lecture-format presentation — 60 minute lecture-format presentation on safer sex and safer injection based on CDC guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). There are no theory-driven active skill building elements oriented towards safer sex or safer injection.
  Other Names: Control
  Arms: Group A

SUMMARY:
The investigators propose a highly efficient four-arm (factorial) trial to simultaneously test the efficacy of two behavioral interventions aimed at:

* increasing condom use in the context of ongoing drug use and
* decreasing needle and paraphernalia sharing

among female sex workers who also inject drugs in two Mexican-U.S. border cities: Tijuana and Ciudad Juarez.

DETAILED DESCRIPTION:
Our specific aims are:

* Aim 1: To evaluate the efficacy of a behavioral intervention to decrease sharing of syringes and injection paraphernalia among FSW-IDUs. We hypothesize that FSW-IDUs in the active experimental injection risk reduction condition will report: (a) less receptive and distributive needle sharing; (b) less sharing of injection paraphernalia; (c) obtaining syringes and injection paraphernalia from safer sources.
* Aim 2: To evaluate the efficacy of a behavioral intervention to increase condom use among FSW-IDUs in the context of ongoing drug use. We hypothesize that FSW-IDUs in the active experimental sexual risk reduction condition will: (a) report less unprotected vaginal and anal sex; and (b) have fewer incident cases of specific STIs.
* Aim 3: To evaluate the joint effects of these two behavioral interventions to increase condom use and reduce sharing of needles and syringes/injection paraphernalia among FSW-IDUs. We hypothesize that the joint effect of these interventions will generate greater risk reductions compared to either intervention alone.
* Aim 4: To determine the extent to which theoretically-important components of our interventions (i.e., self-efficacy, outcome expectancies, attitudes, intentions) represent underlying mechanisms of change in primary outcomes (i.e., sexual- and injection-related risk reductions).
* Aim 5: To explore subgroup differences in the efficacy of: a) the sexual risk reduction, and b) the injection risk reduction intervention based on background characteristics, contextual factors, social factors and intrapersonal factors.

ELIGIBILITY:
Inclusion Criteria:

* be biologically female
* be at least 18 years old
* report having exchanged sex for money, goods or drugs within the last month
* report having injected drugs within the last month
* report having unprotected vaginal or anal sex at least once in last 30 days
* report sharing needles/syringes or other injection paraphernalia (i.e., cottons, cookers, water) at least once in the last month
* live in Tijuana, Ciudad Juarez or its suburbs, as determined through municipal boundaries in each city
* test HIV-negative at baseline
* agree to receive antibiotic treatment for chlamydia, gonorrhea, syphilis trichomonas vaginalis or bacterial vaginosis if they test positive at baseline.

Exclusion Criteria:

If women report:

* consistent use of condoms for vaginal and anal sex with all male partners during the previous month
* not being able to provide verification of injection drug use (i.e. track marks)
* not sharing needles/syringes or paraphernalia at least once in the last month
* being under 18 years of age
* being male or transgender
* being incapable of giving informed consent
* planning to permanently move outside of the municipal boundaries of Tijuana or Ciudad Juarez within the next year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffanie A Strathdee, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- Mexico (2):
  - Sadec-Femap, Ciudad Juárez, Chihuahua
  - PrevenCasa, AC, Tijuana, Estado de Baja California

REFERENCES:
- [Derived] Jain JP, Bristow CC, Pines HA, Harvey-Vera A, Rangel G, Staines H, Patterson TL, Strathdee SA. Factors in the HIV risk environment associated with bacterial vaginosis among HIV-negative female sex workers who inject drugs in the Mexico-United States border region. BMC Public Health. 2018 Aug 20;18(1):1032. doi: 10.1186/s12889-018-5965-9. PMID 30126411
- [Derived] Strathdee SA, Abramovitz D, Lozada R, Martinez G, Rangel MG, Vera A, Staines H, Magis-Rodriguez C, Patterson TL. Reductions in HIV/STI incidence and sharing of injection equipment among female sex workers who inject drugs: results from a randomized controlled trial. PLoS One. 2013 Jun 13;8(6):e65812. doi: 10.1371/journal.pone.0065812. Print 2013. PMID 23785451
- [Derived] Vera A, Abramovitz D, Lozada R, Martinez G, Rangel MG, Staines H, Patterson TL, Strathdee SA. Mujer Mas Segura (Safer Women): a combination prevention intervention to reduce sexual and injection risks among female sex workers who inject drugs. BMC Public Health. 2012 Aug 14;12:653. doi: 10.1186/1471-2458-12-653. PMID 22891807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment took place between October 28, 2008 through May 31, 2010 in Tijuana and November 15, 2008 through July 30, 2010 in Ciudad Juarez.
  Data Collection for this study has been completed and the study is in the analysis phase.
Pre-assignment Details: Targeted sampling techniques were used. Potential participants were approached at venues such as motels, hotels, brothels, shooting galleries, bars, alleys and street corners in both cities. Interested parties were referred to the project offices or a mobile unit for eligibility screening.
Groups:
- A: Didactic Safer Injection & Sexual Activity Education: In each city, 75 women will participate in a 60 minute didactic presentation and printed materials on safer sex and safer injection based on Centers for Disease Control and Prevention (CDC) guidelines for Human Immuno-deficiency Virus (HIV) counseling, testing, and referral and materials from Mexico's National Center for AIDS (Acquired Immuno-Deficiency Syndrome)Studies (CENSIDA).
  In this component, there will be no theory-driven active skill building elements oriented towards safer sex or safer injection.
- B: Interactive Injection Risk & Didactic Safer Sex Education: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] counseling session.
  This one on one intervention incorporates elements of motivational interviewing (MI) and principles of social cognitive theory and theory of reasoned action(SCT/TRA) to address the context of unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared.
  In addition, participants will be provided a lecture-type presentation on safer sex. However, in this component, there will be no theory-driven active skill building elements oriented towards safer sex.
- C:Interactive Sexual Risk & Didactic Safer Injection Eductatio: In each city, 75 women will participate in the 60 minute "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session.
  This one on one intervention incorporates elements of MI and principles of social cognitive theory and theory of reasoned action (SCT/TRA)to address the context of unsafe sex and condom use with clients.
  In addition, participants will be provided a lecture-type presentation on safer injection sharing. However, in this component, there will be no theory-driven active skill building elements oriented towards safer injection behavior.
- D: Interactive Injection & Sexual Risk Intervention: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] and "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session.
  This one-on-one intervention incorporates elements of MI and principles of social cognitive theory and theory of reasoned action (SCT/TRA) to address the context of both, a) unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared; and b) unsafe sex and condom use with clients, and associated risks (e.g., Human Immuno-deficiency Virus (HIV)infection,Sexually Transmitted Infections (STIs, pregnancy).
Period: Overall Study
Arm/Group | A: Didactic Safer Injection & Sexual Activity Education | B: Interactive Injection Risk & Didactic Safer Sex Education | C:Interactive Sexual Risk & Didactic Safer Injection Eductatio | D: Interactive Injection & Sexual Risk Intervention
Started | 144 | 146 | 148 | 146
Completed | 139 (We defined "completed" as having at least one follow-up visit) | 143 (We defined "completed" as having at least one follow-up visit) | 143 (We defined "completed" as having at least one follow-up visit) | 142 (We defined "completed" as having at least one follow-up visit)
Not Completed | 5 | 3 | 5 | 4
Not completed — Death | 2 | 2 | 3 | 3
Not completed — Lost to Follow-up | 3 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- A: Didactic Safer Injection & Sexual Activity Education: In each city, 75 women will participate in a 60 minute lecture-format presentation and printed materials on safer sex and safer injection based on CDC guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). In this component, there will be no theory-driven active skill building elements oriented towards safer sex or safer injection.
- B: Interactive Injection Risk & Didactic Safer Sex Education: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] counseling session. This one on one intervention incorporates elements of motivational interviewing (MI) and principles of SCT/TRA to address the context of unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared. In addition, participants will be provided a didactic presentation on safer sex. However, in this component, there will be no theory-driven active skill building elements oriented towards safer sex.
- C:Interactive Sexual Risk & Didactic Safer Injection Education: In each city, 75 women will participate in the 60 minute "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one on one intervention incorporates elements of motivational interviewing (MI)and principles of social cognitive theory and theory of reasoned action (SCT/TRA) to address the context of unsafe sex and condom use with clients. In addition, participants will be provided a lecture-format presentation on safer injection sharing. However, in this component, there will be no theory-driven active skill building elements oriented towards safer injection behavior.
- D: Interactive Injection & Sexual Risk Intervention: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] and "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one-on-one intervention incorporates elements of motivational interviewing (MI) and principles of Social Cognitive Theory and Theory of Reasoned Action (SCT/TRA) to address the context of both, a) unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared; and b) unsafe sex and condom use with clients, and associated risks (e.g., HIV, STIs, pregnancy).
- Total: Total of all reporting groups
Arm/Group | A: Didactic Safer Injection & Sexual Activity Education | B: Interactive Injection Risk & Didactic Safer Sex Education | C:Interactive Sexual Risk & Didactic Safer Injection Education | D: Interactive Injection & Sexual Risk Intervention | Total
Number analyzed (Participants) | 144 | 146 | 148 | 146 | 584
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 (2742) [27 to 42] | 32 (2740) [27 to 40] | 34 (2740) [29 to 40] | 34 (2940) [28 to 40] | 33 (2740) [27 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 146 | 148 | 146 | 584
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 144 | 146 | 148 | 146 | 584

OUTCOME MEASURES:

1. Primary Outcome: Combined HIV/STI 12-month Incidence Rates of HIV, Syphilis, Chlamydia, Gonorrhea and Trichomonas Vaginalis.
Description: Combined incidence for HIV/STI was calculated over the 12-month study period and included only those who a) had at least one follow-up visit and b) at baseline tested negative for HIV and any of the aforementioned STIs.
  In the calculations we accounted for the time each participant spent at risk of HIV/any STI during the follow-up period, by using available information on each participant for each time point (i.e. baseline, 4-, 8-, and 12-months was used).
  The analytic method used for this outcome analysis was Poisson regression with robust variance estimation. The outcome variable was a binary variable indicating whether a participant has contracted HIV or a new STI during the 12-month follow-up period. The primary factor of interest was the intervention group. The log ("time spent at risk of HIV/any STI") was used as an offset variable in order to account for the time spent at risk of HIV/any STI by each participant.
Time Frame: 12 months, with measuring points at baseline and at 4, 8, and 12 months past baseline
Measure: Number; unit: incidence density per 100 person years
Arm/Group | A: Didactic Safer Injection & Sexual Activity Education | B: Interactive Injection Risk & Didactic Safer Sex Education | C:Interactive Sexual Risk & Didactic Safer Injection Eductatio | D: Interactive Injection & Sexual Risk Intervention
Number analyzed (Participants) | 139 | 143 | 143 | 142
incidence density per 100 person years | 65.02 | 67.66 | 35.02 | 54.04

2. Secondary Outcome: Change (Baseline to 4-, 8-, and 12-months) in the Mean Number of Unprotected Sex Acts With Clients.
Description: The analytic method used for a) was negative binomial regression with the number of unprotected sex acts with clients as the outcome variable and intervention group, time point (baseline, 4-, 8-, and 12-months), and the interaction between the two as the main effects of interest.
Time Frame: 12 months, with measuring points at baseline and at 4, 8, and 12 months past baseline
Population: The data was analyzed by study location. In Tijuana, there were 284 participants (143 in the intervention and 141 in the control group) and in Ciudad Juarez there were 300 participants (151 in the intervention and 149 in the control group).
Measure: Mean (Standard Deviation); unit: Number of unprotected sex acts
Groups:
- Intervention Group (Arm C+Arm D): The intervention group was created by combining Arm C (i.e., interactive sexual risk and didactic safer injection education) and Arm D (i.e., interactive sexual risk and interactive injection risk)
- Control Group (Arm A+Arm B): The control group was created by combining Arm A (i.e., didactic sexual risk and didactic safer injection education) and Arm B (i.e., didactic sexual risk and interactive injection risk).
Arm/Group | Intervention Group (Arm C+Arm D) | Control Group (Arm A+Arm B)
Number analyzed (Participants) | 294 | 290
Number of unprotected sex acts
  Tijuana (Baseline): number analyzed (Participants) | 143 | 141
  Tijuana (Baseline) | 37.91 (46.79) | 34.76 (36.63)
  Tijuana (4-months): number analyzed (Participants) | 143 | 141
  Tijuana (4-months) | 13.83 (25.81) | 11.94 (23.15)
  Tijuana (8-months): number analyzed (Participants) | 143 | 141
  Tijuana (8-months) | 5.27 (16.28) | 5.99 (16.18)
  Tijuana (12-months): number analyzed (Participants) | 143 | 141
  Tijuana (12-months) | 5.60 (14.58) | 5.38 (16.35)
  Ciudad Juarez (Baseline): number analyzed (Participants) | 151 | 149
  Ciudad Juarez (Baseline) | 46.67 (43.48) | 54.10 (94.38)
  Ciudad Juarez (4-months): number analyzed (Participants) | 151 | 149
  Ciudad Juarez (4-months) | 18.63 (25.14) | 24.09 (41.50)
  Ciudad Juarez (8-months): number analyzed (Participants) | 151 | 149
  Ciudad Juarez (8-months) | 15.98 (21.92) | 20.77 (42.23)
  Ciudad Juarez (12-months): number analyzed (Participants) | 151 | 149
  Ciudad Juarez (12-months) | 11.89 (20.29) | 18.76 (26.53)

3. Secondary Outcome: Change (Baseline to 4-, 8-, and 12-months) in the Proportional Odds of Higher Receptive Needle Sharing
Description: For a) we asked: "In the past month, how often have you used a needle or syringe that you knew or suspected had been used before by someone else?" (possible responses: 1=never, 2=sometimes, 3=about half the time, 4=often, 5=always), with a higher response indicating a higher risk. The intervention effect was evaluated by conducting ordinal logistic regression, with the frequency of receptive needle sharing as the outcome variable and Group (Intervention vs. Control), Visit (Baseline, 4-months, 8-months, and 12-months) and the interaction term between the two (Visit*Group) as the main effects. Our primary interest was the Visit*Group interaction, with a significant corresponding p-value being indicative of an intervention effect.
Time Frame: 12 months, with measuring points at baseline and at 4, 8, and 12 months past baseline
Population: Analyses for the secondary outcomes were stratified by site. Of the total 292 participants in the Intervention Group, 142 were in Tijuana and 150 in Cd. Juarez. Similarly, of the 292 participants in the Control Group, 142 were in Tijuana and 150 in Cd Juarez.
Measure: Mean (95% Confidence Interval); unit: Odds Receptive Needle Sharing
Groups:
- Intervention Group (Arm B+Arm D): The Intervention Group was created by combining those who received Arm B (i.e., Interactive Injection Risk & Didactic Safer Sex Education) and Arm D(i.e., Interactive Injection &Sexual Risk Intervention).
- Control Group (Arm A+ Arm C): The Control Group was created by combining Arm A( i.e., those who received the Didactic Safer Injection & Sexual Activity Education) and Arm C (i.e., those who received Interactive Sexual Risk & Didactic Safer Injection Education).
Arm/Group | Intervention Group (Arm B+Arm D) | Control Group (Arm A+ Arm C)
Number analyzed (Participants) | 292 | 292
Odds Receptive Needle Sharing
  Tijuana (Baseline): number analyzed (Participants) | 142 | 142
  Tijuana (Baseline) | 3.01 [2.18 to 4.15] | 2.83 [2.14 to 3.74]
  Tijuana (4 Months): number analyzed (Participants) | 142 | 142
  Tijuana (4 Months) | 0.32 [0.23 to 0.46] | 0.26 [0.18 to 0.38]
  Tijuana (8 Months): number analyzed (Participants) | 142 | 142
  Tijuana (8 Months) | 0.18 [0.12 to 0.27] | 0.16 [0.11 to 0.25]
  Tijuana (12 months): number analyzed (Participants) | 142 | 142
  Tijuana (12 months) | 0.15 [0.10 to 0.23] | 0.13 [0.08 to 0.21]
  Ciudad Juarez (baseline): number analyzed (Participants) | 142 | 150
  Ciudad Juarez (baseline) | 2.45 [1.79 to 3.35] | 1.911 [1.40 to 2.60]
  Ciudad Juarez (4 months): number analyzed (Participants) | 150 | 150
  Ciudad Juarez (4 months) | 0.85 [0.59 to 1.23] | 0.69 [0.47 to 1.02]
  Ciudad Juarez (8 months): number analyzed (Participants) | 150 | 150
  Ciudad Juarez (8 months) | 0.53 [0.37 to 0.77] | 0.71 [0.49 to 1.03]
  Ciudad Juarez (12 months): number analyzed (Participants) | 150 | 150
  Ciudad Juarez (12 months) | 0.38 [0.27 to 0.55] | 0.56 [0.39 to 0.79]
Statistical Analysis 1: Comparison: Intervention Group (Arm B+Arm D) vs Control Group (Arm A+ Arm C); Alternative hypothesis: There is a difference between the intervention and the control group with respect to the change in the odds of higher receptive needle sharing. (i.e., The interaction between study visit (baseline, 4-, 8-, and 12-months) and intervention group will be significant at 0.05 significance level. Over time, the intervention group will experience a significant decline in receptive needle sharing but the control group will not.); Test type: Superiority; p = 0.036, Mixed Models Analysis — P-value is for the Ciudad Juarez site and it corresponds to the interaction between group (Intervention vs. Control) and study visit (12-months vs. baseline); To examine the receptive needle sharing outcome, we used ordinal logistic regression for correlated data via GEE with the correlation matrix estimated empirically from the data. The final analyses were stratified by site. The final ordinal logistic regression models included the following main effects: Group, Visit, and Visit*Group interaction, with our primary interest in the Visit*Group interaction, as a significant p-value would be indicative of an intervention effect

4. Secondary Outcome: Change (Baseline to 4-, 8-, and 12-months) in the Mean Score of the Injection Risk Index (IRI).
Description: The injection risk index (IRI) was calculated by averaging the responses to the following five questions:
  1. In the past month, how often have you used a needle or syringe that you knew or suspected had been used before by someone else?
  2. In the past month, how often was a new syringe used to divide the drug?
  3. In the past month, how often did you use a bottle-cap/spoon/cooker after someone else had used it?
  4. In the past month, how often did you use a cotton filter for a needle after someone else had used it?
  5. In the past month, how often did you use rinse water to clean needles after someone else had used it? The possible responses to the questions were coded as follows: 0=never, 1=sometimes, 2=about half the time, 3=often, 4=always. Before averaging the responses to the five questions, the responses to the second question were reversed coded to yield the same direction as the responses to the other four questions. IRI range: 0-20. Higher IRI-->higher risk.
Time Frame: 12 months, with measuring points at baseline and at 4, 8, and 12 months past baseline
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: IRI Score
Arm/Group | Intervention Group (Arm B+Arm D) | Control Group (Arm A+ Arm C)
Number analyzed (Participants) | 292 | 292
IRI Score
  Tijuana (Baseline): number analyzed (Participants) | 142 | 142
  Tijuana (Baseline) | 3.393 [3.240 to 3.553] | 3.358 [3.203 to 3.520]
  Tijuana (4 Months): number analyzed (Participants) | 142 | 142
  Tijuana (4 Months) | 1.916 [1.723 to 2.131] | 1.855 [1.673 to 2.057]
  Tijuana (8 months) | 1.697 [1.508 to 1.910] | 1.648 [1.474 to 1.844]
  Tijuana (12 months) | 1.551 [1.382 to 1.741] | 1.542 [1.368 to 1.737]
  Ciudad Juarez (baseline): number analyzed (Participants) | 150 | 150
  Ciudad Juarez (baseline) | 3.236 [3.045 to 3.439] | 3.07 [2.889 to 3.267]
  Ciudad Juarez (4 months): number analyzed (Participants) | 150 | 150
  Ciudad Juarez (4 months) | 2.418 [2.200 to 2.658] | 2.362 [2.142 to 2.606]
  Ciudad Juarez (8 months) | 2.146 [1.937 to 2.378] | 2.311 [2.095 to 2.549]
  Ciudad Juarez (12 months) | 1.827 [1.657 to 2.015] | 2.070 [1.879 to 2.282]
Statistical Analysis 1: Comparison: Intervention Group (Arm B+Arm D) vs Control Group (Arm A+ Arm C); Alternative hypothesis: There is a difference between the intervention and the control group with respect to the change in the mean score IRI (i.e., The interaction between study visit (baseline, 4-, 8-, and 12-months) and intervention group will be significant at 0.05 significance level. Over time, the intervention group will experience a significant decline in the IRI but the control group will not.); Test type: Superiority; p = 0.013, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; We used gamma regression for correlated data via GEE, with the correlation matrix estimated empirically from the data. The final analyses were stratified by site. The final gamma regression models included the following main effects: Group, Visit, and Visit*Group interaction, with our primary interest in the Visit*Group interaction, as a significant p-value would be indicative of an intervention effect

ADVERSE EVENTS:
Time Frame: October 2008 through July 2010.
Description: Participant reports; death certificates
Groups:
- A: Didactic Safer Injection and Sexual Activity Education: In each city, 75 women will participate in a 60 minute didactic presentation and printed materials on safer sex and safer injection based on CDC guidelines for HIV counseling, testing, and referral and materials from Mexico's National Center for AIDS Studies (CENSIDA). In this component, there will be no theory-driven active skill building elements oriented towards safer sex or safer injection.
- B: Interactive Injection Risk Intervention and Didactic Safer: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] counseling session. This one on one intervention incorporates elements of motivational interviewing (MI) and principles of SCT/TRA to address the context of unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared. In addition, participants will be provided a didactic presentation on safer sex. However, in this component, there will be no theory-driven active skill building elements oriented towards safer sex.
- C:Interactive Sexual Risk Intervention & Didactic Safer: In each city, 75 women will participate in the 60 minute "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one on one intervention incorporates elements of MI and principles of SCT/TRA to address the context of unsafe sex and condom use with clients. In addition, participants will be provided a didactic presentation on safer injection sharing. However, in this component, there will be no theory-driven active skill building elements oriented towards safer injection behavior.
- D: Interactive Injection and Sexual Risk Intervention: In each city, 75 women will participate in the 60 minute "Di No a las Jeringas Contaminadas" ['Say No to Contaminated Syringes'] and "Di No Al Sexo Inseguro" [Say No to Unsafe Sex'] counseling session. This one-on-one intervention incorporates elements of MI and principles of SCT/TRA to address the context of both, a) unsafe injection sharing and the extent to which syringes and other injection paraphernalia is shared; and b) unsafe sex and condom use with clients, and associated risks (e.g., HIV, STIs, pregnancy).
Arm/Group | A: Didactic Safer Injection and Sexual Activity Education | B: Interactive Injection Risk Intervention and Didactic Safer | C:Interactive Sexual Risk Intervention & Didactic Safer | D: Interactive Injection and Sexual Risk Intervention
Serious Adverse Events (participants affected / at risk) | 5/144 | 3/146 | 8/148 | 4/146
Other Adverse Events (participants affected / at risk) | 0/144 | 0/146 | 0/148 | 0/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Didactic Safer Injection and Sexual Activity Education (N=144) | B: Interactive Injection Risk Intervention and Didactic Safer (N=146) | C:Interactive Sexual Risk Intervention & Didactic Safer (N=148) | D: Interactive Injection and Sexual Risk Intervention (N=146)
Participants Affected/at risk (Social circumstances) | 5 (5) | 3 (3) | 8 (8) | 4 (4) — Deceased and lost to follow up due to circumstances beyond study participation

LIMITATIONS AND CAVEATS:
Observed important site differences at enrollment need to be considered in outcome analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No